CLINICAL TRIAL: NCT06646146
Title: A Single-Center, Prospective, Randomized Controlled Clinical Study on the Efficacy of Autologous Fat Grafting in Improving Hair Transplantation Outcomes for Patients With Localized Scleroderma-Related Alopecia
Brief Title: Study on the Efficacy of Autologous Fat Grafting in Improving Hair Transplantation Outcomes for Patients With Localized Scleroderma-Related Alopecia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC -2024-353
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Fat Grafting; Hair Transplantation; Localized Scleroderma
Keywords: fat grafting; localized scleroderma; alopecia; hair transplantation
MeSH Terms: conditions — Scleroderma, Localized; Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fat Graft Combined with Hair Transplantation Group (Experimental)
  Interventions: Procedure: Fat grafting combine with hair transplantation
- Hair Transplantation Group (Active Comparator)
  Interventions: Procedure: Hair transplantation

INTERVENTIONS:
Procedure: Fat grafting combine with hair transplantation — Patients enrolled in this experiment will be divided into two groups.The experimental group will have autologous fat tissue harvested during surgery for fat grafting in the patient's alopecia area, and a subsequent hair transplantation will be performed after three months when the transplanted fat has stabilized and survived.
  Arms: Fat Graft Combined with Hair Transplantation Group
Procedure: Hair transplantation — Patients enrolled in this experiment will be divided into two groups. The control group will undergo a simple hair transplantation surgery.
  Arms: Hair Transplantation Group

SUMMARY:
Investigating the efficacy and safety of autologous fat grafting combined with hair transplantation for the treatment of hair loss in patients with localized scleroderma."

DETAILED DESCRIPTION:
Localized scleroderma is an autoimmune disorder affecting the connective tissue, with skin fibrosis being the primary symptom, potentially leading to skin hardening, atrophy, and hair loss.For facial deformities associated with localized scleroderma, current treatments primarily involve medication, which can ameliorate disease activity but does not reverse the condition. Hair transplantation can improve alopecia, although the survival rate of hair follicles in patients with scleroderma may be lower than in the general population.

Autologous fat grafting is a plastic surgery technique used for soft tissue augmentation and tissue regeneration. The stem cells and growth factors present in adipose tissue contribute to hair regrowth. Studies have indicated that autologous fat grafting, when used adjunctively with hair transplantation, can enhance the survival rate of hair follicles and increase patient satisfaction.Our research team has developed a patented adipose matrix vascular component known as ECM/SVF-gel. This component is rich in active cells and holds potential for regenerative medicine. It has been widely applied clinically to effectively ameliorate scar fibrosis and promote wound healing.

Based on existing research, we hypothesize that fat grafting may improve hair loss in patients with localized scleroderma and increase the survival rate of hair follicles. We plan to conduct a randomized controlled study comparing hair transplantation assisted by ECM/SVF-gel with traditional hair transplantation to validate our hypothesis and provide a more effective treatment option for patients with scleroderma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with clinical symptoms consistent with localized scleroderma (LoSCAT score can be used to assist in diagnosis).

  2. Diagnosed with secondary alopecia caused by localized scleroderma. 3. A history of hair loss in the affected area for more than 6 months, with an adequate supply of donor hair.

  4. The disease is inactive and has been in a stationary phase for over a year (patients have no ongoing or intermittent hair loss accompanied by local pain, itching, or burning; scalp biopsy indicates no inflammatory cell infiltration, hair follicle orifices have disappeared, and hair follicles are replaced by connective tissue).

  5. The general condition is stable, and the patient can tolerate anesthesia and surgery.

  6. BMI is greater than or equal to 17. 7. Age between 18 and 59. 8. The subject and their family are willing and able to comply with postoperative care and follow-up requirements.

  9. The subject and their family have given informed consent and have signed the informed consent form.

Exclusion Criteria:

1. Hair loss area exceeds one-third of the scalp.
2. Infection of the scalp soft tissue.
3. Suffering from psychiatric disorders, hematologic diseases, immune deficiencies, abnormalities in liver or kidney function, severe hypertension, severe diabetes, and other contraindications for surgery.
4. Women who are pregnant or breastfeeding.
5. BMI is less than 17, making it impossible to obtain sufficient fat.
6. Received new vasodilator or immunosuppressive drug treatment within the past 3 months.
7. Applied topical ointments to the surgical area within the past 2 weeks.
8. Positive for HIV, HBV, HCV, HTLV-1 or -2, or syphilis.
9. Patients with a history of tumor formation in the last 5 years.
10. Patients with a prednisolone intake greater than 10 mg/day. Patients deemed unsuitable for participation in this trial by the investigator's judgment.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Hair follicle survival rate | From enrollment to the end of treatment at 12 months
  Number of follicular units per square centimeter at 12 months post-surgery divided by the number of transplanted follicular units per square centimeter immediately post-surgery, multiplied by 100%.

SECONDARY OUTCOMES:
LoSCAT Score | From enrollment to the end of treatment at 1, 3, 6 and 12 months
  Observe the skin lesion conditions of the treatment area before and after treatment, and assess using the LoSCAT scale at 1, 3, 6, and 12 months post-surgery.
Comprehensive efficacy assessment | From enrollment to the end of treatment at 12 months
  Observe and record the hair growth conditions of patients in both groups after surgery and during the follow-up period, and collect relevant statistical data. A comprehensive evaluation is conducted based on four aspects: the coverage rate of the bald area 12 months after surgery, surgical scars, hair density, and hair growth direction. The medical aesthetic effect is evaluated by physicians: Excellent: The bald area is completely covered, the design line is natural and aesthetically pleasing, with no surgical scars, even hair density, and the growth direction is basically consistent with the original hair growth direction; Good: The coverage area of the bald area is ≥80%, with no obvious surgical scars, and the hair density is basically even; Poor: The coverage area of the bald area is <80%, with residual surgical scars, uneven hair density, and disordered hair growth direction. Aesthetics = Excellent + Good.
Patient satisfaction | From enrollment to the end of treatment at 12 months
  At the 12-month follow-up after surgery, a self-made questionnaire is used to evaluate the satisfaction of patients and their families with the post-treatment hair growth in both groups. The scoring range is 0~100 points, divided into five levels: Very Satisfied (85~100 points, including 85 points), Satisfied (70-85 points, including 70 points), Generally Satisfied (55-70 points, including 55 points), Dissatisfied (40-55 points, including 40 points), Very Dissatisfied (below 40 points). Record the patient satisfaction and calculate the patient satisfaction rate
Quality of life score | From enrollment to the end of treatment at 12 months
  Before the start of treatment and 12 months after surgery, the DLQI questionnaire is used to score the quality of life of patients in both groups, with the score increasing as the patient's quality of life improves
Skin biopsy | From enrollment to the end of treatment at 12 months
  Histological assessment of the degree of inflammation and fibrosis in the hair transplant area is conducted 12 months after surgery.

IPD SHARING:
Plan to Share IPD: No